CLINICAL TRIAL: NCT06595875
Title: Modified Thoracoabdominal Nerve Block With Perichondrial Approach in Laparoscopic Cholecystectomy Surgery: A Prospective, Randomized, Controlled, Double-Blind Study
Brief Title: Modified Thoracoabdominal Nerve Block With Perichondrial Approach in Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, the member of the Department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: m-tapa
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- m-tapa block (Active Comparator)
  Interventions: Other: m-tapa block

INTERVENTIONS:
Other: m-tapa block — Patients in Group M were placed in the supine position. After skin antisepsis with 5% povidone-iodine, a sterile drape was placed. The high-frequency (8-13 MHz) linear ultrasound (USG) probe was covered with a sterile sheath, and the transversus abdominis, internal oblique, and external oblique muscles were identified at the 10th costal margin in the sagittal plane at the costochondral angle. The probe was angled sagittally to visualize the costochondral angle at the edge of the 10th rib and to display the posterior surface of the rib cartilage in the midline. Using an in-plane technique, a 22-gauge, 100-millimeter (mm) Stimuplex A peripheral nerve block needle was advanced cranially, and the needle tip was directed towards the posterior surface of the 10th costal cartilage. After negative aspiration, 20 mL of 0.25% bupivacaine was injected under the lower surface of the costal cartilage. The same procedure was repeated on the opposite side.
  Arms: m-tapa block

SUMMARY:
Our primary objective is to evaluate the postoperative numerical rating scale scores in patients undergoing laparoscopic cholecystectomy with an m-TAPA block. Our secondary objectives are to assess the total amount of rescue analgesia consumed, the time to first rescue analgesia, patient satisfaction, and the occurrence of complications.

DETAILED DESCRIPTION:
Patients aged 18-65 with American Society of Anesthesiologists physical status I-III, undergoing laparoscopic cholecystectomy under general anesthesia, were included in the study. Patients with contraindications to regional anesthesia, impaired consciousness, coagulopathy, those using anticoagulants, those with infection at the procedure site, those with allergies to local anesthetics, pregnant women, and emergency cases were excluded from the study.

The primary outcome measures were the numerical rating scale pain scores (0-10, 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain) at 0, 2, 4, 8, 12, and 24 hours postoperatively. The secondary outcome measures included the total amount of rescue analgesic consumed, the time to first rescue analgesia, the occurrence of complications (such as infection, hematoma formation, and local anesthetic systemic toxicity), and patient satisfaction. The age, gender, weight, height, surgery duration of patients in both groups were recorded. A Likert scale (1 = not satisfied at all, 2 = not satisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied) was used to assess patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* American Society of Anesthesiologists physical status I-III
* Laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* Patients with contraindications to regional anesthesia
* Impaired consciousness
* Coagulopathy
* Using anticoagulants
* Infection at the procedure site
* Allergies to local anesthetics
* Pregnant women
* Emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hours
  Our primary objective is to evaluate the postoperative numerical rating scale scores in patients undergoing laparoscopic cholecystectomy with an m-TAPA block. Numerical rating scale score 0-10 point. 0= Very bad, 10= Vey Good.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No